CLINICAL TRIAL: NCT05713552
Title: Evaluation of ACUVUE® OASYS 1-Day for Astigmatism Contact Lenses With Alternative Lidstock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR-6530
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Results first posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Ocular Physiology

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Test/Control (Experimental): Eligible subjects who are habitual soft contact lens wearers will be randomized into the Test/Control sequence, to wear two different study lenses, one at a time, over two wear periods (test then control) with a washout period of 15 minutes between wears. During each wear period the lenses will be worn bilaterally for at least one hour in-office.
  Interventions: Device: Acuvue Oasys 1 Day for Astigmatism with Legacy lidstock; Device: Acuvue Oasys 1 Day for Astigmatism with Amcor laminated lidstock
- Control/Test (Experimental): Eligible subjects who are habitual soft contact lens wearers will be randomized into the Control/Test sequence, to wear two different study lenses, one at a time, over two wear periods (control then test) with a washout period of 15 minutes between wears. During each wear period the lenses will be worn bilaterally for at least one hour in-office.
  Interventions: Device: Acuvue Oasys 1 Day for Astigmatism with Legacy lidstock; Device: Acuvue Oasys 1 Day for Astigmatism with Amcor laminated lidstock

INTERVENTIONS:
Device: Acuvue Oasys 1 Day for Astigmatism with Legacy lidstock — CONTROL
Device: Acuvue Oasys 1 Day for Astigmatism with Amcor laminated lidstock — TEST

SUMMARY:
This will be a single-visit, randomized, double-masked, bilateral wear, non-dispensing, 2-sequence × 2-period crossover study to evaluate subject reported ocular symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. Be between 18 and 39 years of age (inclusive) at the time of screening.
  4. Habitually wear soft contact lenses (either sphere or toric) in both eyes in a daily reusable or daily disposable wear modality (i.e., not extended wear modality). Habitual wear is defined as a minimum of 6 hours per day, for a minimum of 2 days per week during the past four weeks.
  5. Possess a wearable pair of spectacles that provide correction for distance vision.
  6. Have the spherical component of their vertex-corrected distance refraction within the range +4.00 to -9.00 DS (inclusive) in both eyes.
  7. Have the magnitude of the cylindrical component of their vertex-corrected distance refraction below 3.00 DC (inclusive) in both eyes.
  8. Have best corrected monocular distance VA of 20/30 or better in each eye.

Exclusion Criteria:

* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

The subject must not:

1. Be currently pregnant or lactating.
2. Be diabetic.
3. Be currently using any ocular medications or have an ocular infection of any type.
4. Have any ocular or systemic allergies, disease, infection, or use of medication that might contraindicate or interfere with contact lens wear or otherwise compromise study endpoints, including infectious diseases (e.g., hepatitis, tuberculosis), contagious immunosuppressive disease (e.g., Human Immunodeficiency Virus [HIV]), or history of serious mental illness or seizures. See section 9.1 for additional details regarding systemic medications.
5. Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (e.g., SynergEyes, SoftPerm) within the past 6 months.
6. Be currently wearing monovision or multifocal contact lenses or be currently wearing lenses in an extended wear modality.
7. Have a history of strabismus or amblyopia.
8. Be an employee (e.g., Investigator, Coordinator, Technician) or family member of an employee of investigational clinic.
9. Have participated in a contact lens or lens care product clinical trial within 7 days prior to study enrollment.
10. Have clinically significant (Grade 3 or 4 on the FDA classification scale) slit lamp findings (e.g., corneal edema, neovascularization or staining, tarsal abnormalities or bulbar injection) or other corneal or ocular disease or abnormalities that may contraindicate contact lens wear or otherwise compromise study endpoints (including entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis).
11. Have fluctuations in vision due to clinically significant dry eye or other ocular conditions.
12. Have had or have planned (within the study period) ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.).

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (1):
- VRC, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 31 subjects were enrolled in this study. Of those enrolled, 30 subjects were dispensed at least one study lens, while 1 subject failed to meet all eligibility criteria. Of those dispensed, all 30 subjects completed the study.
Groups:
- Test/Control: Subjects randomized to receive the Test lens during the first period and the Control lens during the second period.
- Control/Test: Subjects randomized to receive the Control lens during the first period and the Test lens during the second period.
Period: Period 1
Arm/Group | Test/Control | Control/Test
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Test/Control | Control/Test
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects dispensed a study lens.
Groups:
- Dispensed Subjects: All subjects dispensed a study lens.
Arm/Group | Dispensed Subjects
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.5 (6.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 9
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 5
  Black or African American | 3
  Native Hawaiian or Other Pacific Islander | 1
  White | 21
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Eyes With Moderate or Severe Subject-Reported Ocular Symptoms
Description: Ocular symptoms were assessed using open-ended question. Investigators asked each subject if they experienced any eye symptoms or problems with lens wear when wearing the study lenses. If responded "Yes", then subject characterized each symptom to the following scale for each eye: 0 = Not Applicable or Not Recorded, 1 = Mild and results in little or no interference with lens wear, 2 = Moderate AND/OR occasionally interferes with lens wear, and 3 = Severe AND/OR frequently interferes with lens wear. Investigators classified each subject reported symptom into these categories: Burning/stinging, Itchiness/Scratchiness, Dryness, Lens Awareness, Grittiness/Foreign Body Sensation, Redness, Irritation/Discomfort, Cloudy/Blurry/Hazy, Variable Vision, and Other. The data was dichotomized across all symptoms, where Y=1 if any "moderate" or "severe" ocular symptoms were reported and Y=0 otherwise. The proportion of eyes with any "moderate" or "severe" ocular symptoms was reported for each lens.
Time Frame: Up to 1-Hour Follow-Up
Population: All subjects that were dispensed at least one study lens.
Measure: Number; unit: Proportion of eyes
Units Other Than Participants: Eyes
Groups:
- Test: Subjects that wore the Test lens during either the first or second period of the study.
- Control: Subjects that wore the Control lens during either the first or second period of the study.
Arm/Group | Test | Control
Number analyzed (Participants) | 30 | 30
Number analyzed (Eyes) | 60 | 60
Proportion of eyes
  15-Minute Follow-up | 0 | 0
  1-Hour Follow-up | 0 | 0

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; approximately 1-day per subject.
Arm/Group | Test | Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/52/NCT05713552/Prot_SAP_000.pdf